CLINICAL TRIAL: NCT02073578
Title: Peroral Endoscopic Myotomy (POEM) for the Treatment of Achalasia
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kyle A Perry, Assistant Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011H0240
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Achalasia
Keywords: achalasia; POEM; peroral endoscopic myotomy; myotomy; Heller myotomy
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): Peroral Endoscopic Myotomy (POEM)
  Interventions: Procedure: Peroral Endoscopic Myotomy (POEM)

INTERVENTIONS:
Procedure: Peroral Endoscopic Myotomy (POEM) — Endoscopy myotomy for treatment of achalasia

SUMMARY:
This is a pilot study for a new endoscopic treatment of achalasia. Up to 25 patients will be recruited for this trial, with the intent to treat 20 patients.

DETAILED DESCRIPTION:
This is a pilot study for a new endoscopic treatment of achalasia. Up to 25 patients will be recruited for this trial, with the intent to treat or attempt to treat 20 patients. Patients for whom a POEM has been attempted but not completed (conversion to open or laparoscopic surgery, POEM surgery aborted and not re-attempted). Patients who proceed to study treatment will undergo ten years of follow-up as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Achalasia
* Age 16-80
* ASA Class 1-3

Exclusion Criteria:

* Pregnancy
* Any prior surgical or endoscopic treatment for achalasia -- first eight subjects.

After eight subjects have been treated as part of this study, this exclusion criteria no longer applies

* Patients who are taking immunosuppressive medications or are immunocompromised
* Patients on anticoagulant medications or abnormal coagulation tests
* Patients with severe medical comorbidities, in the judgment of the treating surgeon

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of POEM Procedure | Intraoperative to one year follow-up
  To assess adverse events related to POEM
Long-term patient-reported quality of life | Baseline to one year follow-up
  To assess change in quality of life from baseline, based on validated quality of life measures, at baseline through 1 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Perry, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States